CLINICAL TRIAL: NCT04414930
Title: Pharmacologic Augmentation of Targeted Cognitive Training in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Neal R. Swerdlow, M.D., Ph.D., Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R33MH123603-01 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects complete 30 sessions of Targeted Cognitive Training (2-3 times per week), and receive placebo po 1 hour prior to each training.
  Interventions: Drug: Placebo
- Active Drug (Active Comparator): Subjects complete 30 sessions of Targeted Cognitive Training (2-3 times per week), and receive amphetamine 5 mg po 1 hour prior to each training.
  Interventions: Drug: d-amphetamine

INTERVENTIONS:
Drug: d-amphetamine — Subjects complete 30 sessions of Targeted Cognitive Training (2-3 times per week), and receive amphetamine 5 mg po 1 hour prior to each training.
  Arms: Active Drug
Drug: Placebo — Subjects complete 30 sessions of Targeted Cognitive Training (2-3 times per week), and receive placebo po 1 hour prior to each training.
  Arms: Placebo

SUMMARY:
These studies look to conduct efficient pilot testing of a novel intervention strategy for chronic psychotic disorders - Pharmacologic Augmentation of Cognitive Therapy (PACT) - via an experimental medicine approach. Antipsychotics are the major therapeutic tool for chronic psychotic disorders, including schizophrenia, but do not significantly alter their course or real-life impact. Specific cognitive therapies achieve modest symptom reduction and improved function and cognition in psychosis patients, including "bottom-up" sensory-based targeted cognitive training (TCT). While benefits of TCT are evident at the group level, almost half of all patients demonstrate little or no cognitive gains after 30-40 hours (h) of TCT. For patients and clinicians, the costs and logistical complexities associated with these time- and resource-intensive interventions can be prohibitive. We propose and will test a novel "augmentation strategy" for using medications to specifically enhance the benefits of TCT in schizophrenia.

DETAILED DESCRIPTION:
Subjects who meet criteria for study entry come to UCSD where consenting and a comprehensive screening and diagnostic assessment including a Mini-International Neuropsychiatric Interview are conducted. After initial screening, subjects return twice, approximately 7 days apart, for biomarker assessment after challenge with placebo (PBO) (Test 1) or amphetamine 5 mg po (AMPH) (Test 2). Subjects then enter the "treatment phase", completing up to 30 one-hour targeted cognitive training (TCT) sessions. Subjects are randomized to one of 2 groups: "AMPH Group" receive AMPH (5 mg po) 1h before each TCT session; "PBO Group" receive PBO dosed identically to AMPH. Pill identity (AMPH vs. PBO) is blind to subjects and staff.

TCT sessions are scheduled approximately 3 times each week for 10 weeks. TCT consists of 7 computerized exercises delivered on standardized laptops and headphones. Collectively, these exercises target learning mechanisms involving auditory perception and processing speed (Sound Sweeps, Fine Tuning) and auditory memory (Syllable Stacks, Memory Grid, To-Do List Training, Rhythm Recall, Hear-Hear). Training is structured into blocks that deliver stimulus sets with varying temporal and psychophysical parameters to allow continuous learning and improvement. Blocks consist of 10-35 adaptive trials where the subject's progression depends on their performance. Exercises apply an n-up/m-down algorithm to responses to estimate psychophysical thresholds while ensuring that participants remain engaged and challenged at an appropriate level (~80% accuracy) as their abilities improve.

Clinical and functional outcome measures are acquired at "baseline", and 1-2 days after completion of 10, 20 and 30 TCT sessions and 12 weeks post-training. Urine toxicology screens and Columbia Suicide Severity Rating Scales are performed at least weekly, prior to a TCT session. A treatment satisfaction scale (100 mm line) rates expectations at the start of the study and actual experience of treatment in three areas: "satisfaction", "hard work" and "worthwhile." Subjects from both groups return to UCSD 12 weeks after the TCT has ended, and outcome measures are reassessed to test the "durability" of benefits.

ELIGIBILITY:
Inclusion criteria include:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder, depressed type
* Written informed consent to participate in the study
* Age 18 - 55
* Absence of dementia or mental retardation
* Urine toxicology negative for recreational drugs
* Fluent and literate in English (needed for completion of WIN and QuickSIN)

Exclusion criteria include:

* Meets DSM-IV criteria for current substance abuse or dependence and has been substance abstinent for less than 30 days
* A history of traumatic brain injury
* Auditory or visual impairments severe enough to prevent study participation
* Under conservatorship (determined by Anasazi)
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal R Serdlow, M.D., Ph.D., Principal Investigator — UC San Diego
Locations (1):
- Clinical Teaching Facility (CTF-B102) at UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Antipsychotic-medicated outpatients with a primary diagnosis of SZ or schizoaffective disorder (depressed type) ages 18-55 were recruited from the San Diego community between 11/9/2020 and 3/13/2024. Of the 68 consented/enrolled participants, 28 met inclusion criteria and were randomized to treatment.
Pre-assignment Details: A total of 68 participants were enrolled but 35 were excluded for not meeting inclusion criteria and 5 withdrew from the study. Therefore 28 participants were randomized.
Groups:
- Amphetamine: Subjects complete 30 sessions of Targeted Cognitive Training (2-3 times per week), and receive amphetamine 5 mg po 1 hour prior to each training.
  d-amphetamine: Subjects complete 30 sessions of Targeted Cognitive Training (2-3 times per week), and receive amphetamine 5 mg po 1 hour prior to each training.
Period: Overall Study
Arm/Group | Placebo | Amphetamine
Started | 10 | 18
Completed | 9 | 15
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drug | Total
Number analyzed (Participants) | 10 | 18 | 28
Age, Continuous [Mean (Full Range); unit: years] | 41.7 [32 to 54] | 46.7 [34 to 59] | 44.9 [32 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 6 | 13 | 19
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 2 | 9 | 11
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 18 | 28

OUTCOME MEASURES:

1. Primary Outcome: Primary Clinical Outcome PANSS Total Score (PANSSt)
Description: Positive & Negative Symptom Scale total (PANSSt) PANSS Total Score is the primary clinical outcome measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks).
  The PANSS total score has a range 30-210, with higher scores indicating worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 65.4 (5.7) | 55.6 (3.2)
  Post-10 | 67.1 (4.6) | 49.8 (3.1)
  Post-20 | 61.0 (5.7) | 50.5 (2.5)
  Post-30 | 60.1 (7.3) | 46.5 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measures ANOVA; p = 0.28, ANOVA — The threshold for statistical significance was p<0.05; Repeated measure ANOVA group x time

2. Primary Outcome: Primary Functional Outcome WHODAS
Description: Primary World Health Organization Disability Schedule (WHODAS 2.0) Function will be assessed via the World Health Organization Disability Schedule 2.0 (WHODAS 2.0) at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The WHODAS 2.0 has a range 12-60, with higher scores indicating worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 26.6 (4.7) | 53.1 (8.0)
  Post-10 | 38.1 (9.4) | 43.7 (7.2)
  Post-20 | 29.6 (6.8) | 34.5 (8.7)
  Post-30 | 34.7 (8.9) | 32.1 (4.8)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.05, ANOVA — The threshold for statistical significance was p<0.05; Repeated measure ANOVA group x time

3. Primary Outcome: Primary Neurocognitive Outcome MCCB-C
Description: MATRICS Consensus Cognitive Battery Global Composite T-score (MCCB-C) The MCCB Global Composite T-score (MCCB-C) is the primary neurocognitive outcome measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The MATRICS Consensus Cognitive Battery (MCCB) composite T-score has no minimum or maximum score because it uses T-scores, which are standardized based on a community sample. A normal range MCCB composite T-score is between 40 and 60 and higher scores indicate better neurocognitive outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 17.7 (3.2) | 29.8 (5.0)
  Post-10 | 19.3 (4.9) | 30.4 (5.1)
  Post-20 | 21.3 (3.8) | 34.3 (4.6)
  Post-30 | 20.3 (4.7) | 30.5 (4.8)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.93, ANOVA — The threshold for significance was p<0.05

4. Secondary Outcome: Secondary Clinical Outcome Measure PANSSp
Description: Positive & Negative Symptom Scale positive symptom subscale (PANSSp) measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The PANSSp is rated with 1 to 7 points ranging from absent to extreme. The range is 7-49 and higher scores indicate worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 16.6 (2.3) | 15.2 (1.3)
  Post-10 | 16.6 (2.0) | 12.5 (1.0)
  Post-20 | 16.0 (1.9) | 13.9 (1.1)
  Post-30 | 14.7 (1.9) | 11.8 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.43, ANOVA — The threshold for significance was p<0.05; Repeated measure ANOVA group x time

5. Secondary Outcome: Secondary Clinical Outcome Measure PANSSn
Description: Positive & Negative Symptom Scale negative symptom subscale (PANSSn)measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The PANSSn is rated with 1 to 7 points ranging from absent to extreme. The range is 7-49 and higher scores indicate worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 16.6 (2.1) | 12.8 (1.1)
  Post-10 | 17.4 (1.4) | 12.9 (1.3)
  Post-20 | 15.9 (2.6) | 12.1 (0.7)
  Post-30 | 17.4 (3.1) | 12.0 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.77, ANOVA — The threshold for significance was p<0.05; Repeated measure ANOVA group x time

6. Secondary Outcome: Psychotic Symptoms PSYRATS Hallucinations
Description: Psychotic Symptom Rating Scales (PSYRATS hallucination subscale) assesses auditory hallucinations measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The PSYRATS auditory hallucinations subscale (AHS) consisting of 11 items, with each item being rated from 0 (absent) to 4 (severe), range 0-44, with higher scores indicating more severe auditory hallucinations or worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 2.7 (1.8) | 16.3 (2.8)
  Post-10 | 3.4 (3.4) | 11.3 (2.9)
  Post-20 | 5.6 (2.9) | 13.9 (2.7)
  Post-30 | 0.0 (0.0) | 10.4 (3.1)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.50, ANOVA — The threshold for significance is p<0.05; Repeated measure ANOVA group x time

7. Secondary Outcome: Manic Symptoms YMRS
Description: Young Mania Rating Scale total score measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The range for the YMRS total score is 0-60, with higher scores indicating more severe manic symptoms or worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 7.0 (2.1) | 5.6 (1.4)
  Post-10 | 6.0 (1.4) | 2.6 (1.0)
  Post-20 | 5.9 (2.1) | 3.3 (1.0)
  Post-30 | 6.0 (1.9) | 2.5 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.636, ANOVA — The threshold for significance is p<0.05; Repeated measure ANOVA group x time

8. Secondary Outcome: Current Depressive Symptoms PHQ
Description: Patient Health Questionnaire-9 (PHQ-9) total score measured at baseline vs. post-TCT session 10, 20 and 30 (approximately 10 weeks). The PHQ-9 has a range from 0 to 27 with higher scores indicating more severe depression or worse outcome.
Time Frame: approximately 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Amphetamine
Number analyzed (Participants) | 10 | 18
score on a scale
  Baseline | 4.4 (1.4) | 6.3 (1.7)
  Post-10 | 6.3 (1.7) | 2.9 (0.9)
  Post-20 | 4.0 (1.3) | 4.4 (1.9)
  Post-30 | 3.9 (2.1) | 3.9 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Amphetamine; Test type: Superiority — Repeated measure ANOVA; p = 0.19, ANOVA — The threshold for significance was p<0.05; Repeated measure ANOVA group x time

ADVERSE EVENTS:
Time Frame: Data was collected over the course of the study participation, about 10 weeks
Description: Gastrointestinal symptoms (e.g. bloating, diarrhea, cramps) were all assessed/monitored under the general description "gastrointestinal symptoms".
Arm/Group | Placebo | Amphetamine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 7/10 | 10/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Amphetamine (N=18)
increase in psychiatric symptoms (Psychiatric disorders) | 3 | 4 — Increased psychiatric symptoms including increased auditory hallucinations and worse mood
Gastrointestinal (Gastrointestinal disorders) | 2 | 3 — Gastrointestinal symptoms (e.g. bloating, diarrhea, cramps)
Restless night (Psychiatric disorders) | 1 | 3 — Restless Night (1 night)
Worsening TD-related tremor (Nervous system disorders) | 1 | 0 — Worsening Tardive Dyskinesia-related tremor
Minor Accident (e.g. trip, fall) (General disorders) | 1 | 1 — Minor Accident (e.g. trip, fall)
Elevated blood pressure and/or heart rate (Cardiac disorders) | 1 | 2 — Elevated blood pressure and/or heart rate as measured at study visit
ear ache (Ear and labyrinth disorders) | 1 | 0 — ear ache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04414930/Prot_001.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04414930/SAP_002.pdf
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT04414930/ICF_000.pdf